CLINICAL TRIAL: NCT03694704
Title: Study of Auditory Performance on Postoperative Prosodic Tests in Subjects Implanted With a MED-EL Cochlear Implant and Using a FineHearing Strategy. Prospective Longitudinal Multicentric Study
Brief Title: Study of Auditory Performance on Prosodic Tests in Cochlear Implanted Subjects Using a Fine Structure Strategy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MED-EL_FS_prosody_french_study
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2022-05

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant; stimulation strategy; sound coding strategy
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CI with FineHearing Strategy (Experimental): cochlear implant with FineHearing strategy
  Interventions: Device: FineHearing strategy

INTERVENTIONS:
Device: FineHearing strategy — Cochlear implant with FineHearing strategy

SUMMARY:
Main objective:

Investigate how the FineHearing strategy of the MED-EL cochlear implant can extract prosody based solely on the frequency of the voice fundamental (F0) in speech

Secondary objectives:

Evaluate the time evolution of the results of prosodic tests Evaluate the time evolution of the results of differential frequency threshold test Evaluate the time evolution of vocal audiometric tests in silence and noise Evaluate the correlation between prosodic test results and frequency differential threshold results

DETAILED DESCRIPTION:
Introduction:

Prosodie is the study of the phenomena of accentuation and intonation (variation of pitch, duration and intensity) allowing the conveyance of information related to the sense such as the relief, but also the assertion, interrogation, injunction, exclamation ...

It has a role at the grammatical, emotional and pragmatic levels of communication by informing about the emotional state of the speaker (sad / happy), about sex and identity, about the type of statement (question / affirmation) and about the borders in the sentences.

The auditory cues that play a role in the perception of prosody include changes in the fundamental frequency F0 (ie vibrational frequency of the speaker's vocal cords) during a speech, the duration of the syllables, or the rate or intensity of the speech. [Di Christo 2013] The cochlear implant is a device for auditory rehabilitation. Its principle is to transform the analog signals recorded by a microphone into digital signals that directly stimulate the fibers of the auditory nerve through electrodes inserted into the cochlea. [HAS 2012, HAS 2007, http://www.has-sante.fr] Cochlear implants are indicated in cases of severe or profound sensorineural deafness.

Conventional stimulation strategies in cochlear implants (e.g. ACE, CIS) use the place of the electrode to code the frequency by sending low frequency information on the apical electrodes and high frequency information on the basal electrodes. The stimulation rate of the electrodes is constant. [Wilson & Dorman 2008] The pitch is only partially transmitted by these conventional strategies [Moore 2003; Oxenham 2008] which would explain the poor results of cochlear implants in the perception of music [Bruns & al. 2016; Galvin III & al. 2009; Veekmans & al. 2009; Cooper & al. 2008] and prosody [Kalathottukaren & al. 2015 ; Meister et al. 2011; Meister et al. 2009].

In the FineHearing strategy of the MED-EL implant, the rate of stimulation on the low-frequency electrodes is related to the frequency of the sound and makes it possible to code the frequency information temporally.

[Rader & al. 2016] have studied the contribution of adding to the tonotopic coding of the frequency (classical strategy) a temporal coding of the information by varying the stimulation rate. The results obtained show that providing this frequency information by time coding makes it possible to obtain perceived pitch much closer to the expected pitch (of normal-hearing) and less variability, especially at low frequencies. With fixed stimulation rate (classical strategy) low frequencies are poorly coded, whereas with the variable stimulation rate they are better coded.

The FineHearing coding strategy of MED-EL with long insertion of electrode could therefore make it possible to better transmit the prosody and specifically to better extract the fundamental frequency F0 of the voice.

Objective of the study The objective of the study is to evaluate if the FineHearing strategy of the MED-EL implant allows to better transmit the prosody and specifically by the fundamental frequency of the voice (F0).

Main objective:

Show that the MED-EL FineHearing strategy (with deep insertion of the electrode) allows to extract prosody cues based only on the fundamental frequency F0.

Secondary objectives:

* evaluate differential frequency thresholds and correlation with prosodic performance
* Evaluate the positioning of the electrode array and its effect on prosodic performance

Plan of study:

It is a prospective open multicenter longitudinal study: measures will be done on the patient at 6 and 12 month post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with MED-EL cochlear implant (Sonnet / Synchrony)
* Adult patient (≥ 18 years old) speaking French
* Patient having an estimate of the optimal size of the electrode for its cochlea with the MED-EL software before their implantation.
* Patient with post-implant audiometry thresholds without cochlear implant > 80 dB HL on 250 Hz, 500 Hz and 1000 Hz frequencies (no residual hearing)
* Patient with vocal audiometry in quiet on Fournier's disyllabic words ≥ 70% at 6 months post-activation

Exclusion criteria:

* Retro-cochlear pathology: auditory neuropathy, vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Prosodic test | at 12 month post-activation
  Two versions, question and statement, of each of 12 sentences were recorded. The final 24 stimuli were constructed so that members of a question/statement pair were acoustically identical until the final syllable leaving pitch as the only salient cue for discrimination. the 24 sentences were presented in random order to the patient and he has to say if it is a question or a statement. Each good answer is scored 1 yielding a total between 0 and 24

SECONDARY OUTCOMES:
Differential frequency threshold | at 6 month post-activation
  This test aimed to determine the smallest perceptible difference in F0 between two stimuli for various baseline values of F0. An adaptive procedure is used.
Prosodic test | at 6 month post-activation
  Two versions, question and statement, of each of 12 sentences were recorded. The final 24 stimuli were constructed so that members of a question/statement pair were acoustically identical until the final syllable leaving pitch as the only salient cue for discrimination. the 24 sentences were presented in random order to the patient and he has to say if it is a question or a statement. Each good answer is scored 1 yielding a total between 0 and 24
Vocal audiometry in quiet and noise | at 6 month post-activation
  Word recognition test in quiet with 10 words. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
  Signal to noise ratio (SRT50) to have 50% of sentence recognition in noise. Measure of the speech reception threshold (i.e. the speech intensity in dB SPL) for 50% (SRT50) of comprehension of sentences free field with the cochlear implant.
Differential frequency threshold | at 12 month post-activation
  This test aimed to determine the smallest perceptible difference in F0 between two stimuli for various baseline values of F0. An adaptive procedure is used.
Vocal audiometry in quiet and noise | at 12 month post-activation
  Word recognition test in quiet with 10 words. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
  Signal to noise ratio (SRT50) to have 50% of sentence recognition in noise. Measure of the speech reception threshold (i.e. the speech intensity in dB SPL) for 50% (SRT50) of comprehension of sentences free field with the cochlear implant.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No